CLINICAL TRIAL: NCT01960790
Title: Humira® 40mg Syringe 0.8mL Subcutaneous Injection Special Investigation in Patients With Intestinal Behcet's Disease
Brief Title: Special Investigation in Patients With Intestinal Behcet's Disease (All Case Investigation)
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P14-152
Record Dates: First submitted 2013-07-16; First posted 2013-10-11 (Estimated); Results first posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2018-05

CONDITIONS: Behcet's Disease
Keywords: Humira®; Behcet's Disease; Adalimumab
MeSH Terms: conditions — Behcet Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Participants who received Humira®: Humira® 40 mg (marketed product) every other week (eow) for subcutaneous injection after initial dosage of 160 mg and 2nd dosage of 80 mg in two weeks after the initial administration

SUMMARY:
This investigation was conducted to obtain the following information regarding the use of Adalimumab (Humira®) 40mg Syringe 0.8mL for Subcutaneous Injection in patients with Intestinal Behcet's Disease.

1. Incidence and conditions of occurrence of adverse reactions in clinical practice
2. Factors likely to affect the safety and effectiveness

ELIGIBILITY:
Inclusion Criteria:

* All patients who received Adalimumab for the treatment of Intestinal Behcet's disease (not sufficiently responsive to existing therapies, e.g. steroids, immunomodulator)

Exclusion Criteria:

Contraindications according to the Package Insert include patients who had any of the following:

* serious infections
* tuberculosis
* a history of hypersensitivity to any ingredient of Humira®
* demyelinating disease or a history of demyelinating disease
* congestive cardiac failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants who received Humira® (Adalimumab) for the treatment of Intestinal Behcet's disease
Sampling Method: Non-Probability Sample
Enrollment: 473 (Actual)
Dates: Start 2013-05-25; Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Osamu Mikami, MD, Study Director — AbbVie

REFERENCES:
- [Derived] Suzuki Y, Hagiwara T, Kobayashi M, Morita K, Shimamoto T, Hibi T. Long-term safety and effectiveness of adalimumab in 462 patients with intestinal Behcet's disease: results from a large real-world observational study. Intest Res. 2021 Jul;19(3):301-312. doi: 10.5217/ir.2020.00013. Epub 2020 Aug 20. PMID 32814420
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 473 participants were enrolled in the study; 462 participants were analyzed for safety and 383 participants were analyzed for efficacy.
Period: Overall Study
Arm/Group | Participants Who Received Humira®
Started | 473
Completed | 462
Not Completed | 11
Not completed — Survey forms could not be recovered | 3
Not completed — Treat with Humira outside survey period | 3
Not completed — Transferred to another hospital | 4
Not completed — Unevaluable for safety | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population: all enrolled participants who received at least 1 dose of study drug
Arm/Group | Participants Who Received Humira®
Number analyzed (Participants) | 462
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Demographic data was unavailable for one participant.
  years
    number analyzed (Participants) | 461
    (all) | 46.3 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Demographic data was unavailable for one participant.
  Participants
    number analyzed (Participants) | 461
    Female | 225
    Male | 236
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 461
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reactions
Description: The number of participants with adverse drug reactions with evaluation beginning upon administration of Humira® is assessed.
Time Frame: Up to Week 156
Population: Safety analysis set: All participants who received at least one administration of Humira® during the study (after informed consent or first administration of Humira®) and for 70 days following the last scheduled administration of Humira®.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received Humira®
Number analyzed (Participants) | 462
Participants
  Infections and infestations | 47
  Neoplasms benign, malignant and unspecified | 5
  Blood and lymphatic system disorders | 6
  Immune system disorders | 1
  Endocrine disorders | 3
  Metabolism and nutrition disorders | 1
  Psychiatric disorders | 3
  Nervous system disorders | 7
  Eye disorders | 1
  Vascular disorders | 5
  Respiratory, thoracic and mediastinal disorders | 9
  Gastrointestinal Disorders | 20
  Hepatobiliary disorders | 4
  Skin and subcutaneous tissue disorder | 6
  Musculoskeletal and connective tissue disorder | 9
  Pregnancy, puerperium and perinatal conditions | 1
  General disorders and adminstration site condition | 19
  Investigations | 22
  Injury, poisoning and procedural complications | 1

2. Secondary Outcome: Global Assessment of Gastrointestinal Symptoms
Description: Study participants completed a global assessment of their gastrointestinal symptoms on a 5-grade scale. Assessment is graded from 0 to 4: 0=free of symptoms; 1=symptoms existed since the last visit, but did not affect participant's daily life; 2=symptoms existed since the last visit and slightly affected participant's daily life; 3=symptoms existed since the last visit and affected participant's daily life; 4=symptoms existed since the last visit and critically affected participant's daily life.
Time Frame: Up to Week 156
Population: All participants who received Humira® to treat gastro-intestinal Behcet's disease and were evaluable for efficacy.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received Humira®
Number analyzed (Participants) | 383
Participants
  Baseline: number analyzed (Participants) | 369
  Baseline: Global assessment score = 0 | 52
  Baseline: Global assessment score = 1 | 55
  Baseline: Global assessment score = 2 | 76
  Baseline: Global assessment score = 3 | 88
  Baseline: Global assessment score = 4 | 98
  Week 4: number analyzed (Participants) | 323
  Week 4: Global assessment score = 0 | 153
  Week 4: Global assessment score = 1 | 85
  Week 4: Global assessment score = 2 | 44
  Week 4: Global assessment score = 3 | 33
  Week 4: Global assessment score = 4 | 8
  Week 8: number analyzed (Participants) | 315
  Week 8: Global assessment score = 0 | 176
  Week 8: Global assessment score = 1 | 72
  Week 8: Global assessment score = 2 | 38
  Week 8: Global assessment score = 3 | 19
  Week 8: Global assessment score = 4 | 10
  Week 12: number analyzed (Participants) | 292
  Week 12: Global assessment score = 0 | 169
  Week 12: Global assessment score = 1 | 72
  Week 12: Global assessment score = 2 | 32
  Week 12: Global assessment score = 3 | 12
  Week 12: Global assessment score = 4 | 7
  Week 24: number analyzed (Participants) | 240
  Week 24: Global assessment score = 0 | 152
  Week 24: Global assessment score = 1 | 44
  Week 24: Global assessment score = 2 | 34
  Week 24: Global assessment score = 3 | 8
  Week 24: Global assessment score = 4 | 2
  Week 52: number analyzed (Participants) | 221
  Week 52: Global assessment score = 0 | 142
  Week 52: Global assessment score = 1 | 45
  Week 52: Global assessment score = 2 | 22
  Week 52: Global assessment score = 3 | 10
  Week 52: Global assessment score = 4 | 2
  Week 76: number analyzed (Participants) | 176
  Week 76: Global assessment score = 0 | 112
  Week 76: Global assessment score = 1 | 38
  Week 76: Global assessment score = 2 | 18
  Week 76: Global assessment score = 3 | 8
  Week 76: Global assessment score = 4 | 0
  Week 104: number analyzed (Participants) | 172
  Week 104: Global assessment score = 0 | 113
  Week 104: Global assessment score = 1 | 39
  Week 104: Global assessment score = 2 | 17
  Week 104: Global assessment score = 3 | 3
  Week 104: Global assessment score = 4 | 0
  Week 128: number analyzed (Participants) | 50
  Week 128: Global assessment score = 0 | 29
  Week 128: Global assessment score = 1 | 12
  Week 128: Global assessment score = 2 | 8
  Week 128: Global assessment score = 3 | 0
  Week 128: Global assessment score = 4 | 1
  Week 156: number analyzed (Participants) | 49
  Week 156: Global assessment score = 0 | 32
  Week 156: Global assessment score = 1 | 8
  Week 156: Global assessment score = 2 | 9
  Week 156: Global assessment score = 3 | 0
  Week 156: Global assessment score = 4 | 0

3. Secondary Outcome: Global Assessment of Gastrointestinal Symptoms of Behcet's Disease
Description: Study participants completed a global assessment of their gastrointestinal symptoms (including abdominal pain, diarrhea and other gastrointestinal symptoms such as abdominal distension, abdominal tenderness, and hemorrhage) on a 5-grade scale. Assessment is graded from 0 to 4: 0=free of symptoms; 1=symptoms existed since the last visit, but did not affect participant's daily life; 2=symptoms existed since the last visit and slightly affected participant's daily life; 3=symptoms existed since the last visit and affected participant's daily life; 4=symptoms existed since the last visit and critically affected participant's daily life.
Time Frame: Up to Week 156
Population: All participants who received Humira® to treat gastro-intestinal Behcet's disease and were evaluable for efficacy.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received Humira®
Number analyzed (Participants) | 368
Participants
  Abdominal pain at week 0 (baseline): Global assessment score = 0 | 89
  Abdominal pain at week 0 (baseline): Global assessment score = 1 | 56
  Abdominal pain at week 0 (baseline): Global assessment score = 2 | 74
  Abdominal pain at week 0 (baseline): Global assessment score = 3 | 82
  Abdominal pain at week 0 (baseline): Global assessment score = 4 | 67
  Abdominal pain at week 4: number analyzed (Participants) | 322
  Abdominal pain at week 4: Global assessment score = 0 | 181
  Abdominal pain at week 4: Global assessment score = 1 | 69
  Abdominal pain at week 4: Global assessment score = 2 | 39
  Abdominal pain at week 4: Global assessment score = 3 | 27
  Abdominal pain at week 4: Global assessment score = 4 | 6
  Abdominal pain at week 8: number analyzed (Participants) | 314
  Abdominal pain at week 8: Global assessment score = 0 | 202
  Abdominal pain at week 8: Global assessment score = 1 | 59
  Abdominal pain at week 8: Global assessment score = 2 | 28
  Abdominal pain at week 8: Global assessment score = 3 | 20
  Abdominal pain at week 8: Global assessment score = 4 | 5
  Abdominal pain at week 12: number analyzed (Participants) | 292
  Abdominal pain at week 12: Global assessment score = 0 | 193
  Abdominal pain at week 12: Global assessment score = 1 | 54
  Abdominal pain at week 12: Global assessment score = 2 | 26
  Abdominal pain at week 12: Global assessment score = 3 | 13
  Abdominal pain at week 12: Global assessment score = 4 | 6
  Abdominal pain at week 24: number analyzed (Participants) | 239
  Abdominal pain at week 24: Global assessment score = 0 | 174
  Abdominal pain at week 24: Global assessment score = 1 | 28
  Abdominal pain at week 24: Global assessment score = 2 | 29
  Abdominal pain at week 24: Global assessment score = 3 | 6
  Abdominal pain at week 24: Global assessment score = 4 | 2
  Abdominal pain at week 52: number analyzed (Participants) | 220
  Abdominal pain at week 52: Global assessment score = 0 | 158
  Abdominal pain at week 52: Global assessment score = 1 | 31
  Abdominal pain at week 52: Global assessment score = 2 | 21
  Abdominal pain at week 52: Global assessment score = 3 | 10
  Abdominal pain at week 52: Global assessment score = 4 | 0
  Abdominal pain at week 76: number analyzed (Participants) | 177
  Abdominal pain at week 76: Global assessment score = 0 | 129
  Abdominal pain at week 76: Global assessment score = 1 | 26
  Abdominal pain at week 76: Global assessment score = 2 | 14
  Abdominal pain at week 76: Global assessment score = 3 | 8
  Abdominal pain at week 76: Global assessment score = 4 | 0
  Abdominal pain at week 104: number analyzed (Participants) | 173
  Abdominal pain at week 104: Global assessment score = 0 | 132
  Abdominal pain at week 104: Global assessment score = 1 | 31
  Abdominal pain at week 104: Global assessment score = 2 | 8
  Abdominal pain at week 104: Global assessment score = 3 | 2
  Abdominal pain at week 104: Global assessment score = 4 | 0
  Abdominal pain at week 128: number analyzed (Participants) | 50
  Abdominal pain at week 128: Global assessment score = 0 | 36
  Abdominal pain at week 128: Global assessment score = 1 | 8
  Abdominal pain at week 128: Global assessment score = 2 | 4
  Abdominal pain at week 128: Global assessment score = 3 | 1
  Abdominal pain at week 128: Global assessment score = 4 | 1
  Abdominal pain at week 156: number analyzed (Participants) | 49
  Abdominal pain at week 156: Global assessment score = 0 | 36
  Abdominal pain at week 156: Global assessment score = 1 | 5
  Abdominal pain at week 156: Global assessment score = 2 | 8
  Abdominal pain at week 156: Global assessment score = 3 | 0
  Abdominal pain at week 156: Global assessment score = 4 | 0
  Diarrhoea at week 0 (baseline): Global assessment score = 0 | 167
  Diarrhoea at week 0 (baseline): Global assessment score = 1 | 61
  Diarrhoea at week 0 (baseline): Global assessment score = 2 | 54
  Diarrhoea at week 0 (baseline): Global assessment score = 3 | 50
  Diarrhoea at week 0 (baseline): Global assessment score = 4 | 36
  Diarrhoea at week 4: number analyzed (Participants) | 322
  Diarrhoea at week 4: Global assessment score = 0 | 226
  Diarrhoea at week 4: Global assessment score = 1 | 52
  Diarrhoea at week 4: Global assessment score = 2 | 27
  Diarrhoea at week 4: Global assessment score = 3 | 14
  Diarrhoea at week 4: Global assessment score = 4 | 3
  Diarrhoea at week 8: number analyzed (Participants) | 314
  Diarrhoea at week 8: Global assessment score = 0 | 232
  Diarrhoea at week 8: Global assessment score = 1 | 54
  Diarrhoea at week 8: Global assessment score = 2 | 18
  Diarrhoea at week 8: Global assessment score = 3 | 7
  Diarrhoea at week 8: Global assessment score = 4 | 3
  Diarrhoea at week 12: number analyzed (Participants) | 292
  Diarrhoea at week 12: Global assessment score = 0 | 221
  Diarrhoea at week 12: Global assessment score = 1 | 37
  Diarrhoea at week 12: Global assessment score = 2 | 26
  Diarrhoea at week 12: Global assessment score = 3 | 5
  Diarrhoea at week 12: Global assessment score = 4 | 3
  Diarrhoea at week 24: number analyzed (Participants) | 239
  Diarrhoea at week 24: Global assessment score = 0 | 181
  Diarrhoea at week 24: Global assessment score = 1 | 35
  Diarrhoea at week 24: Global assessment score = 2 | 21
  Diarrhoea at week 24: Global assessment score = 3 | 2
  Diarrhoea at week 24: Global assessment score = 4 | 0
  Diarrhoea at week 52: number analyzed (Participants) | 220
  Diarrhoea at week 52: Global assessment score = 0 | 176
  Diarrhoea at week 52: Global assessment score = 1 | 28
  Diarrhoea at week 52: Global assessment score = 2 | 12
  Diarrhoea at week 52: Global assessment score = 3 | 4
  Diarrhoea at week 52: Global assessment score = 4 | 0
  Diarrhoea at week 76: number analyzed (Participants) | 177
  Diarrhoea at week 76: Global assessment score = 0 | 131
  Diarrhoea at week 76: Global assessment score = 1 | 31
  Diarrhoea at week 76: Global assessment score = 2 | 10
  Diarrhoea at week 76: Global assessment score = 3 | 5
  Diarrhoea at week 76: Global assessment score = 4 | 0
  Diarrhoea at week 104: number analyzed (Participants) | 173
  Diarrhoea at week 104: Global assessment score = 0 | 135
  Diarrhoea at week 104: Global assessment score = 1 | 26
  Diarrhoea at week 104: Global assessment score = 2 | 10
  Diarrhoea at week 104: Global assessment score = 3 | 2
  Diarrhoea at week 104: Global assessment score = 4 | 0
  Diarrhoea at week 128: number analyzed (Participants) | 50
  Diarrhoea at week 128: Global assessment score = 0 | 36
  Diarrhoea at week 128: Global assessment score = 1 | 11
  Diarrhoea at week 128: Global assessment score = 2 | 3
  Diarrhoea at week 128: Global assessment score = 3 | 0
  Diarrhoea at week 128: Global assessment score = 4 | 0
  Diarrhoea at week 156: number analyzed (Participants) | 49
  Diarrhoea at week 156: Global assessment score = 0 | 37
  Diarrhoea at week 156: Global assessment score = 1 | 8
  Diarrhoea at week 156: Global assessment score = 2 | 4
  Diarrhoea at week 156: Global assessment score = 3 | 0
  Diarrhoea at week 156: Global assessment score = 4 | 0
  Other gastrointestinal symptoms at week 0/baseline: Global assessment score = 0 | 124
  Other gastrointestinal symptoms at week 0/baseline: Global assessment score = 1 | 54
  Other gastrointestinal symptoms at week 0/baseline: Global assessment score = 2 | 61
  Other gastrointestinal symptoms at week 0/baseline: Global assessment score = 3 | 68
  Other gastrointestinal symptoms at week 0/baseline: Global assessment score = 4 | 61
  Other gastrointestinal symptoms at week 4: number analyzed (Participants) | 322
  Other gastrointestinal symptoms at week 4: Global assessment score = 0 | 219
  Other gastrointestinal symptoms at week 4: Global assessment score = 1 | 49
  Other gastrointestinal symptoms at week 4: Global assessment score = 2 | 31
  Other gastrointestinal symptoms at week 4: Global assessment score = 3 | 16
  Other gastrointestinal symptoms at week 4: Global assessment score = 4 | 7
  Other gastrointestinal symptoms at week 8: number analyzed (Participants) | 314
  Other gastrointestinal symptoms at week 8: Global assessment score = 0 | 226
  Other gastrointestinal symptoms at week 8: Global assessment score = 1 | 44
  Other gastrointestinal symptoms at week 8: Global assessment score = 2 | 27
  Other gastrointestinal symptoms at week 8: Global assessment score = 3 | 10
  Other gastrointestinal symptoms at week 8: Global assessment score = 4 | 7
  Other gastrointestinal symptoms at week 12: number analyzed (Participants) | 292
  Other gastrointestinal symptoms at week 12: Global assessment score = 0 | 220
  Other gastrointestinal symptoms at week 12: Global assessment score = 1 | 40
  Other gastrointestinal symptoms at week 12: Global assessment score = 2 | 21
  Other gastrointestinal symptoms at week 12: Global assessment score = 3 | 7
  Other gastrointestinal symptoms at week 12: Global assessment score = 4 | 4
  Other gastrointestinal symptoms at week 24: number analyzed (Participants) | 239
  Other gastrointestinal symptoms at week 24: Global assessment score = 0 | 188
  Other gastrointestinal symptoms at week 24: Global assessment score = 1 | 28
  Other gastrointestinal symptoms at week 24: Global assessment score = 2 | 19
  Other gastrointestinal symptoms at week 24: Global assessment score = 3 | 2
  Other gastrointestinal symptoms at week 24: Global assessment score = 4 | 2
  Other gastrointestinal symptoms at week 52: number analyzed (Participants) | 220
  Other gastrointestinal symptoms at week 52: Global assessment score = 0 | 172
  Other gastrointestinal symptoms at week 52: Global assessment score = 1 | 26
  Other gastrointestinal symptoms at week 52: Global assessment score = 2 | 15
  Other gastrointestinal symptoms at week 52: Global assessment score = 3 | 6
  Other gastrointestinal symptoms at week 52: Global assessment score = 4 | 1
  Other gastrointestinal symptoms at week 76: number analyzed (Participants) | 177
  Other gastrointestinal symptoms at week 76: Global assessment score = 0 | 138
  Other gastrointestinal symptoms at week 76: Global assessment score = 1 | 20
  Other gastrointestinal symptoms at week 76: Global assessment score = 2 | 13
  Other gastrointestinal symptoms at week 76: Global assessment score = 3 | 5
  Other gastrointestinal symptoms at week 76: Global assessment score = 4 | 1
  Other gastrointestinal symptoms at week 104: number analyzed (Participants) | 173
  Other gastrointestinal symptoms at week 104: Global assessment score = 0 | 143
  Other gastrointestinal symptoms at week 104: Global assessment score = 1 | 17
  Other gastrointestinal symptoms at week 104: Global assessment score = 2 | 10
  Other gastrointestinal symptoms at week 104: Global assessment score = 3 | 3
  Other gastrointestinal symptoms at week 104: Global assessment score = 4 | 0
  Other gastrointestinal symptoms at week 128: number analyzed (Participants) | 50
  Other gastrointestinal symptoms at week 128: Global assessment score = 0 | 36
  Other gastrointestinal symptoms at week 128: Global assessment score = 1 | 11
  Other gastrointestinal symptoms at week 128: Global assessment score = 2 | 1
  Other gastrointestinal symptoms at week 128: Global assessment score = 3 | 1
  Other gastrointestinal symptoms at week 128: Global assessment score = 4 | 1
  Other gastrointestinal symptoms at week 156: number analyzed (Participants) | 49
  Other gastrointestinal symptoms at week 156: Global assessment score = 0 | 37
  Other gastrointestinal symptoms at week 156: Global assessment score = 1 | 7
  Other gastrointestinal symptoms at week 156: Global assessment score = 2 | 4
  Other gastrointestinal symptoms at week 156: Global assessment score = 3 | 1
  Other gastrointestinal symptoms at week 156: Global assessment score = 4 | 0

4. Secondary Outcome: Number of Participants With Cardinal Symptoms of Behcet's Disease
Description: The presence or absence of symptoms including recurrent aphthous ulcers of oral mucosa, cutaneous symptoms, eye symptoms and ulceration of vulva was assessed at weeks 52, 104 and 156 against presence or absence at baseline.
Time Frame: Up to Week 156
Population: All participants who received Humira® to treat gastro-intestinal Behcet's disease and were evaluable for efficacy.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received Humira®
Number analyzed (Participants) | 220
Participants
  Recurrent aphthous ulcers of oral mucosa at week52: number analyzed (Participants) | 219
  Recurrent aphthous ulcers of oral mucosa at week52: Assessment absence and baseline absence | 99
  Recurrent aphthous ulcers of oral mucosa at week52: Assessment absence and baseline presence | 84
  Recurrent aphthous ulcers of oral mucosa at week52: Assessment presence and baseline absence | 7
  Recurrent aphthous ulcers of oral mucosa at week52: Assessment presence and baseline presence | 29
  Recurrent aphthous ulcer of oral mucosa at week104: number analyzed (Participants) | 172
  Recurrent aphthous ulcer of oral mucosa at week104: Assessment absence and baseline absence | 74
  Recurrent aphthous ulcer of oral mucosa at week104: Assessment absence and baseline presence | 59
  Recurrent aphthous ulcer of oral mucosa at week104: Assessment presence and baseline absence | 13
  Recurrent aphthous ulcer of oral mucosa at week104: Assessment presence and baseline presence | 26
  Recurrent aphthous ulcer of oral mucosa at week156: number analyzed (Participants) | 49
  Recurrent aphthous ulcer of oral mucosa at week156: Assessment absence and baseline absence | 27
  Recurrent aphthous ulcer of oral mucosa at week156: Assessment absence and baseline presence | 12
  Recurrent aphthous ulcer of oral mucosa at week156: Assessment presence and baseline absence | 5
  Recurrent aphthous ulcer of oral mucosa at week156: Assessment presence and baseline presence | 5
  Cutaneous symptoms at week 52: number analyzed (Participants) | 219
  Cutaneous symptoms at week 52: Assessment absence and baseline absence | 147
  Cutaneous symptoms at week 52: Assessment absence and baseline presence | 56
  Cutaneous symptoms at week 52: Assessment presence and baseline absence | 5
  Cutaneous symptoms at week 52: Assessment presence and baseline presence | 11
  Cutaneous symptoms at week 104: number analyzed (Participants) | 173
  Cutaneous symptoms at week 104: Assessment absence and baseline absence | 123
  Cutaneous symptoms at week 104: Assessment absence and baseline presence | 34
  Cutaneous symptoms at week 104: Assessment presence and baseline absence | 7
  Cutaneous symptoms at week 104: Assessment presence and baseline presence | 9
  Cutaneous symptoms at week 156: number analyzed (Participants) | 49
  Cutaneous symptoms at week 156: Assessment absence and baseline absence | 32
  Cutaneous symptoms at week 156: Assessment absence and baseline presence | 13
  Cutaneous symptoms at week 156: Assessment presence and baseline absence | 4
  Cutaneous symptoms at week 156: Assessment presence and baseline presence | 0
  Eye symptoms at week 52: Assessment absence and baseline absence | 216
  Eye symptoms at week 52: Assessment absence and baseline presence | 3
  Eye symptoms at week 52: Assessment presence and baseline absence | 0
  Eye symptoms at week 52: Assessment presence and baseline presence | 1
  Eye symptoms at week 104: number analyzed (Participants) | 173
  Eye symptoms at week 104: Assessment absence and baseline absence | 168
  Eye symptoms at week 104: Assessment absence and baseline presence | 4
  Eye symptoms at week 104: Assessment presence and baseline absence | 1
  Eye symptoms at week 104: Assessment presence and baseline presence | 0
  Eye symptoms at week 156: number analyzed (Participants) | 49
  Eye symptoms at week 156: Assessment absence and baseline absence | 48
  Eye symptoms at week 156: Assessment absence and baseline presence | 1
  Eye symptoms at week 156: Assessment presence and baseline absence | 0
  Eye symptoms at week 156: Assessment presence and baseline presence | 0
  Ulceration of vulva at week 52: Assessment absence and baseline absence | 184
  Ulceration of vulva at week 52: Assessment absence and baseline presence | 27
  Ulceration of vulva at week 52: Assessment presence and baseline absence | 1
  Ulceration of vulva at week 52: Assessment presence and baseline presence | 8
  Ulceration of vulva at week 104: number analyzed (Participants) | 173
  Ulceration of vulva at week 104: Assessment absence and baseline absence | 151
  Ulceration of vulva at week 104: Assessment absence and baseline presence | 14
  Ulceration of vulva at week 104: Assessment presence and baseline absence | 4
  Ulceration of vulva at week 104: Assessment presence and baseline presence | 4
  Ulceration of vulva at week 156: number analyzed (Participants) | 49
  Ulceration of vulva at week 156: Assessment absence and baseline absence | 42
  Ulceration of vulva at week 156: Assessment absence and baseline presence | 5
  Ulceration of vulva at week 156: Assessment presence and baseline absence | 1
  Ulceration of vulva at week 156: Assessment presence and baseline presence | 1

5. Secondary Outcome: Number of Participants With Accessory Symptoms of Behcet's Disease
Description: The presence or absence of symptoms including arthritis without deformity or stiffness, epididymitis, vascular lesions and moderate to severe central nervous system (CNS) lesions was assessed at weeks 52, 104 and 156 against presence or absence at baseline.
Time Frame: Up to Week 156
Population: All participants who received Humira® to treat gastro-intestinal Behcet's disease and were evaluable for efficacy.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received Humira®
Number analyzed (Participants) | 221
Participants
  Arthritis without deformity/ stiffness at week 52: Assessment absence and baseline absence | 150
  Arthritis without deformity/ stiffness at week 52: Assessment absence and baseline presence | 39
  Arthritis without deformity/ stiffness at week 52: Assessment presence and baseline absence | 11
  Arthritis without deformity/ stiffness at week 52: Assessment presence and baseline presence | 21
  Arthritis without deformity/ stiffness at week 104: number analyzed (Participants) | 174
  Arthritis without deformity/ stiffness at week 104: Assessment absence and baseline absence | 115
  Arthritis without deformity/ stiffness at week 104: Assessment absence and baseline presence | 36
  Arthritis without deformity/ stiffness at week 104: Assessment presence and baseline absence | 14
  Arthritis without deformity/ stiffness at week 104: Assessment presence and baseline presence | 9
  Arthritis without deformity/ stiffness at week 156: number analyzed (Participants) | 49
  Arthritis without deformity/ stiffness at week 156: Assessment absence and baseline absence | 30
  Arthritis without deformity/ stiffness at week 156: Assessment absence and baseline presence | 14
  Arthritis without deformity/ stiffness at week 156: Assessment presence and baseline absence | 5
  Arthritis without deformity/ stiffness at week 156: Assessment presence and baseline presence | 0
  Epididymitis at week 52: Assessment absence and baseline absence | 219
  Epididymitis at week 52: Assessment absence and baseline presence | 0
  Epididymitis at week 52: Assessment presence and baseline absence | 0
  Epididymitis at week 52: Assessment presence and baseline presence | 2
  Epididymitis at week 104: number analyzed (Participants) | 174
  Epididymitis at week 104: Assessment absence and baseline absence | 172
  Epididymitis at week 104: Assessment absence and baseline presence | 2
  Epididymitis at week 104: Assessment presence and baseline absence | 0
  Epididymitis at week 104: Assessment presence and baseline presence | 0
  Epididymitis at week 156: number analyzed (Participants) | 49
  Epididymitis at week 156: Assessment absence and baseline absence | 46
  Epididymitis at week 156: Assessment absence and baseline presence | 1
  Epididymitis at week 156: Assessment presence and baseline absence | 1
  Epididymitis at week 156: Assessment presence and baseline presence | 1
  Vascular lesions at week 52: Assessment absence and baseline absence | 213
  Vascular lesions at week 52: Assessment absence and baseline presence | 0
  Vascular lesions at week 52: Assessment presence and baseline absence | 1
  Vascular lesions at week 52: Assessment presence and baseline presence | 7
  Vascular lesions at week 104: number analyzed (Participants) | 174
  Vascular lesions at week 104: Assessment absence and baseline absence | 168
  Vascular lesions at week 104: Assessment absence and baseline presence | 4
  Vascular lesions at week 104: Assessment presence and baseline absence | 0
  Vascular lesions at week 104: Assessment presence and baseline presence | 2
  Vascular lesions at week 156: number analyzed (Participants) | 49
  Vascular lesions at week 156: Assessment absence and baseline absence | 47
  Vascular lesions at week 156: Assessment absence and baseline presence | 1
  Vascular lesions at week 156: Assessment presence and baseline absence | 1
  Vascular lesions at week 156: Assessment presence and baseline presence | 0
  Moderate to severe CNS lesions at week 52: Assessment absence and baseline absence | 217
  Moderate to severe CNS lesions at week 52: Assessment absence and baseline presence | 1
  Moderate to severe CNS lesions at week 52: Assessment presence and baseline absence | 1
  Moderate to severe CNS lesions at week 52: Assessment presence and baseline presence | 2
  Moderate to severe CNS lesions at week 104: number analyzed (Participants) | 174
  Moderate to severe CNS lesions at week 104: Assessment absence and baseline absence | 171
  Moderate to severe CNS lesions at week 104: Assessment absence and baseline presence | 1
  Moderate to severe CNS lesions at week 104: Assessment presence and baseline absence | 0
  Moderate to severe CNS lesions at week 104: Assessment presence and baseline presence | 2
  Moderate to severe CNS lesions at week 156: number analyzed (Participants) | 49
  Moderate to severe CNS lesions at week 156: Assessment absence and baseline absence | 48
  Moderate to severe CNS lesions at week 156: Assessment absence and baseline presence | 0
  Moderate to severe CNS lesions at week 156: Assessment presence and baseline absence | 1
  Moderate to severe CNS lesions at week 156: Assessment presence and baseline presence | 0

6. Secondary Outcome: Number of Participants With Degree of Improvement of Endoscopic Findings
Description: The number of participants with improvement in endoscopic findings is assessed.
Time Frame: Up to Week 156
Population: All participants who received Humira® to treat gastro-intestinal Behcet's disease and were evaluable for efficacy.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received Humira®
Number analyzed (Participants) | 383
Participants
  Baseline to < Week 24: number analyzed (Participants) | 137
  Baseline to < Week 24: Cured or scarring | 64
  Baseline to < Week 24: Diminished in size | 38
  Baseline to < Week 24: Unchanged | 24
  Baseline to < Week 24: Aggravated | 9
  Baseline to < Week 24: Unassessable | 2
  Week 24 to < Week 52: number analyzed (Participants) | 128
  Week 24 to < Week 52: Cured or scarring | 73
  Week 24 to < Week 52: Diminished in size | 29
  Week 24 to < Week 52: Unchanged | 12
  Week 24 to < Week 52: Aggravated | 6
  Week 24 to < Week 52: Unassessable | 8
  Week 52 to < Week 76: number analyzed (Participants) | 60
  Week 52 to < Week 76: Cured or scarring | 42
  Week 52 to < Week 76: Diminished in size | 6
  Week 52 to < Week 76: Unchanged | 9
  Week 52 to < Week 76: Aggravated | 0
  Week 52 to < Week 76: Unassessable | 3
  Week 76 to < Week 104: number analyzed (Participants) | 49
  Week 76 to < Week 104: Cured or scarring | 29
  Week 76 to < Week 104: Diminished in size | 6
  Week 76 to < Week 104: Unchanged | 7
  Week 76 to < Week 104: Aggravated | 5
  Week 76 to < Week 104: Unassessable | 2
  Week 104 to < Week 128: number analyzed (Participants) | 22
  Week 104 to < Week 128: Cured or scarring | 16
  Week 104 to < Week 128: Diminished in size | 3
  Week 104 to < Week 128: Unchanged | 1
  Week 104 to < Week 128: Aggravated | 1
  Week 104 to < Week 128: Unassessable | 1
  Week 128 to < Week 160: number analyzed (Participants) | 11
  Week 128 to < Week 160: Cured or scarring | 9
  Week 128 to < Week 160: Diminished in size | 1
  Week 128 to < Week 160: Unchanged | 0
  Week 128 to < Week 160: Aggravated | 0
  Week 128 to < Week 160: Unassessable | 1

7. Secondary Outcome: Changes in C-reactive Protein (CRP)
Description: The change in CRP from baseline through the end of the study was assessed.
Time Frame: Up to Week 156
Population: All participants who received Humira® to treat gastro-intestinal Behcet's disease and were evaluable for efficacy.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Participants Who Received Humira®
Number analyzed (Participants) | 383
mg/dL
  Baseline | 2.0239 (3.4242)
  Week 24: number analyzed (Participants) | 231
  Week 24 | 0.5389 (1.5150)
  Week 52: number analyzed (Participants) | 206
  Week 52 | 0.5504 (1.4651)
  Week 76: number analyzed (Participants) | 164
  Week 76 | 0.3348 (0.8126)
  Week 104: number analyzed (Participants) | 161
  Week 104 | 0.4031 (1.1279)
  Week 128: number analyzed (Participants) | 42
  Week 128 | 0.5034 (2.5356)
  Week 156: number analyzed (Participants) | 43
  Week 156 | 0.2246 (0.5808)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from first dose of study drug until 70 days after the last dose of study drug (up to 156 weeks); Serious Adverse Events were collected from the time informed consent was obtained (156 weeks).
Arm/Group | Participants Who Received Humira®
All-Cause Mortality (participants affected / at risk) | 4/462
Serious Adverse Events (participants affected / at risk) | 75/462
Other Adverse Events (participants affected / at risk) | 165/462
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Who Received Humira® (N=462)
BRONCHITIS (Infections and infestations) | 1 (1)
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 1 (1)
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 1 (1)
MENINGITIS LISTERIA (Infections and infestations) | 1 (1)
PERIODONTITIS (Infections and infestations) | 1 (1)
PHARYNGITIS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 5 (5)
PSEUDOMEMBRANOUS COLITIS (Infections and infestations) | 1 (1)
PULMONARY TUBERCULOSIS (Infections and infestations) | 1 (1)
SEPSIS (Infections and infestations) | 3 (3)
ANAL ABSCESS (Infections and infestations) | 1 (1)
INTERVERTEBRAL DISCITIS (Infections and infestations) | 1 (1)
ABDOMINAL ABSCESS (Infections and infestations) | 1 (1)
PNEUMONIA BACTERIAL (Infections and infestations) | 1 (1)
COLONIC ABSCESS (Infections and infestations) | 1 (1)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 2 (2)
VARICELLA ZOSTER VIRUS INFECTION (Infections and infestations) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CHRONIC MYELOMONOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
GASTROINTESTINAL STROMAL TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
MYELODYSPLASTIC SYNDROME TRANSFORMATION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
EPSTEIN-BARR VIRUS ASSOCIATED LYMPHOPROLIFERATIVE DISORDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
ANAEMIA MEGALOBLASTIC (Blood and lymphatic system disorders) | 1 (1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 1 (1)
ADRENAL DISORDER (Endocrine disorders) | 1 (1)
DIABETES INSIPIDUS (Endocrine disorders) | 1 (1)
THYROIDITIS SUBACUTE (Endocrine disorders) | 1 (1)
COMPLETED SUICIDE (Psychiatric disorders) | 1 (1)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1)
BEHCET'S SYNDROME (Vascular disorders) | 11 (11)
SHOCK HAEMORRHAGIC (Vascular disorders) | 1 (1)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2 (2)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
ENTEROCOLITIS (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
ILEAL PERFORATION (Gastrointestinal disorders) | 2 (2)
ILEAL ULCER (Gastrointestinal disorders) | 2 (2)
ILEUS (Gastrointestinal disorders) | 2 (2)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 3 (3)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 2 (2)
PANCREATITIS (Gastrointestinal disorders) | 1 (1)
SMALL INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1)
STOMATITIS (Gastrointestinal disorders) | 1 (1)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
FISTULA OF SMALL INTESTINE (Gastrointestinal disorders) | 1 (1)
DENTAL CYST (Gastrointestinal disorders) | 1 (1)
BILE DUCT STONE (Hepatobiliary disorders) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 2 (2)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1)
FISTULA (Musculoskeletal and connective tissue disorders) | 1 (1)
LUPUS-LIKE SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1)
ABORTION MISSED (Pregnancy, puerperium and perinatal conditions) | 1 (1)
PYREXIA (General disorders) | 7 (7)
C-REACTIVE PROTEIN INCREASED (Investigations) | 2 (2)
PLATELET COUNT DECREASED (Investigations) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 2 (2)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1 (1)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Who Received Humira® (N=462)
ANGULAR CHEILITIS (Infections and infestations) | 1 (1)
BRONCHITIS (Infections and infestations) | 3 (3)
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 2 (2)
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1)
CYSTITIS (Infections and infestations) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 2 (2)
HERPES ZOSTER (Infections and infestations) | 2 (2)
INFLUENZA (Infections and infestations) | 2 (2)
MENINGITIS LISTERIA (Infections and infestations) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 10 (10)
ORAL CANDIDIASIS (Infections and infestations) | 2 (2)
OTITIS MEDIA (Infections and infestations) | 2 (2)
OTITIS MEDIA CHRONIC (Infections and infestations) | 1 (1)
PERIODONTITIS (Infections and infestations) | 1 (1)
PHARYNGITIS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 7 (7)
PSEUDOMEMBRANOUS COLITIS (Infections and infestations) | 1 (1)
PULMONARY TUBERCULOSIS (Infections and infestations) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 1 (1)
SEPSIS (Infections and infestations) | 3 (3)
SINUSITIS (Infections and infestations) | 1 (1)
TINEA PEDIS (Infections and infestations) | 1 (1)
TONSILLITIS (Infections and infestations) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2)
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 2 (2)
ANAL ABSCESS (Infections and infestations) | 3 (3)
ENTERITIS INFECTIOUS (Infections and infestations) | 1 (1)
INTERVERTEBRAL DISCITIS (Infections and infestations) | 1 (1)
ABDOMINAL ABSCESS (Infections and infestations) | 1 (1)
PNEUMONIA BACTERIAL (Infections and infestations) | 2 (2)
LUNG INFECTION (Infections and infestations) | 1 (1)
ENTEROCOLITIS VIRAL (Infections and infestations) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1)
LATENT TUBERCULOSIS (Infections and infestations) | 2 (2)
ORAL HERPES (Infections and infestations) | 1 (1)
COLONIC ABSCESS (Infections and infestations) | 1 (1)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 2 (2)
VARICELLA ZOSTER VIRUS INFECTION (Infections and infestations) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CHRONIC MYELOMONOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
GASTROINTESTINAL STROMAL TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
MYELODYSPLASTIC SYNDROME TRANSFORMATION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
EPSTEIN-BARR VIRUS ASSOCIATED LYMPHOPROLIFERATIVE DISORDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
ANAEMIA (Blood and lymphatic system disorders) | 3 (3)
ANAEMIA MEGALOBLASTIC (Blood and lymphatic system disorders) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
LYMPHADENITIS (Blood and lymphatic system disorders) | 1 (1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 1 (1)
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 1 (1)
SEASONAL ALLERGY (Immune system disorders) | 1 (1)
ADRENAL DISORDER (Endocrine disorders) | 1 (1)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 (1)
DIABETES INSIPIDUS (Endocrine disorders) | 2 (2)
THYROIDITIS SUBACUTE (Endocrine disorders) | 1 (1)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 1 (1)
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2)
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERAMYLASAEMIA (Metabolism and nutrition disorders) | 1 (1)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 (2)
HYPERLIPASAEMIA (Metabolism and nutrition disorders) | 1 (1)
COMPLETED SUICIDE (Psychiatric disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 3 (3)
OBSESSIVE-COMPULSIVE DISORDER (Psychiatric disorders) | 1 (1)
DEPRESSIVE SYMPTOM (Psychiatric disorders) | 1 (1)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 1 (1)
DYSLALIA (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 4 (4)
HYPOAESTHESIA (Nervous system disorders) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 1 (1)
TREMOR (Nervous system disorders) | 1 (1)
CONJUNCTIVITIS ALLERGIC (Eye disorders) | 1 (1)
VITREOUS FLOATERS (Eye disorders) | 1 (1)
ARTERIOSCLEROSIS (Vascular disorders) | 1 (1)
BEHCET'S SYNDROME (Vascular disorders) | 15 (15)
HYPOTENSION (Vascular disorders) | 1 (1)
SHOCK HAEMORRHAGIC (Vascular disorders) | 1 (1)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PHARYNGEAL ULCERATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2 (2)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
UPPER RESPIRATORY TRACT INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 4 (4)
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 3 (3)
DIARRHOEA (Gastrointestinal disorders) | 2 (2)
ENTEROCOLITIS (Gastrointestinal disorders) | 2 (2)
GASTRITIS ALCOHOLIC (Gastrointestinal disorders) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 (3)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 (1)
ILEAL PERFORATION (Gastrointestinal disorders) | 2 (2)
ILEAL ULCER (Gastrointestinal disorders) | 2 (2)
ILEUS (Gastrointestinal disorders) | 2 (2)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 3 (3)
INTESTINAL STENOSIS (Gastrointestinal disorders) | 1 (1)
INTESTINAL ULCER (Gastrointestinal disorders) | 1 (1)
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 1 (1)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 2 (2)
PANCREATITIS (Gastrointestinal disorders) | 1 (1)
SMALL INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1)
STOMATITIS (Gastrointestinal disorders) | 5 (5)
VOMITING (Gastrointestinal disorders) | 3 (3)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 1 (1)
FISTULA OF SMALL INTESTINE (Gastrointestinal disorders) | 1 (1)
FAECES SOFT (Gastrointestinal disorders) | 1 (1)
DENTAL CYST (Gastrointestinal disorders) | 1 (1)
ALCOHOLIC LIVER DISEASE (Hepatobiliary disorders) | 1 (1)
BILE DUCT STONE (Hepatobiliary disorders) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 2 (2)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 2 (2)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 (1)
LIVER DISORDER (Hepatobiliary disorders) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1)
ABORTION MISSED (Pregnancy, puerperium and perinatal conditions) | 1 (1)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 (1)
ASTHENIA (General disorders) | 1 (1)
INJECTION SITE ERYTHEMA (General disorders) | 1 (1)
INJECTION SITE REACTION (General disorders) | 4 (4)
MALAISE (General disorders) | 5 (5)
PAIN (General disorders) | 1 (1)
PYREXIA (General disorders) | 13 (13)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
C-REACTIVE PROTEIN INCREASED (Investigations) | 12 (12)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 2 (2)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 5 (5)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 2 (2)
ANTITHROMBIN III DECREASED (Investigations) | 1 (1)
BLOOD BETA-D-GLUCAN INCREASED (Investigations) | 2 (2)
BRAIN NATRIURETIC PEPTIDE INCREASED (Investigations) | 1 (1)
TRANSAMINASES INCREASED (Investigations) | 1 (1)
COMPUTERISED TOMOGRAM THORAX ABNORMAL (Investigations) | 2 (2)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1)
LIVER FUNCTION TEST INCREASED (Investigations) | 1 (1)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 (6)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
FISTULA (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
LUPUS-LIKE SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1)
DERMAL CYST (Skin and subcutaneous tissue disorders) | 1 (1)
DYSHIDROTIC ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1)
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 1 (1)
HAEMORRHAGE SUBCUTANEOUS (Skin and subcutaneous tissue disorders) | 1 (1)
PRURIGO (Skin and subcutaneous tissue disorders) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 2 (2)
GENERALISED ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1)
DERMATITIS PSORIASIFORM (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2013-06-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT01960790/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT01960790/SAP_001.pdf